CLINICAL TRIAL: NCT03107884
Title: Metformin to Prevent Inactivity-induced Loss of Muscle Health During Aging
Brief Title: Role of Metformin on Muscle Health of Older Adults
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Micah Drummond, Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 93579
Record Dates: First submitted 2017-03-22; First posted 2017-04-11 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Muscle Atrophy; Insulin Resistance
Keywords: Insulin Resistance; Muscle Atrophy; Metformin; Muscle Loss; Inactivity-induced muscle loss; older adults
MeSH Terms: conditions — Muscular Atrophy; Insulin Resistance | interventions — Metformin; Bed Rest

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: drug and placebo will be encapsulated therefore concealing the participant, investigator and outcome assessor to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Metformin (Bed Rest) (Experimental): Metformin will be given to participants incrementally during a 2 week run in period such that they will receive the clinical dose (2 grams per day). During bed rest, participants will be given 1 gram of metformin two times a day (morning and evening). This dosage and frequency will occur during four consecutive days of bed rest.
  Interventions: Drug: Metformin (Bed Rest)
- Placebo (Bed Rest) (Placebo Comparator): Placebo will be given to participants incrementally during a 2 week run in period such that they will receive the same amount of pills as the experimental group. During bed rest, participants will be given the same amount of pills and given at the same time of day (morning and evening) as the experimental group. This strategy will occur during four consecutive days of bed rest.
  Interventions: Drug: Placebo (Bed Rest)
- Metformin (2 week run-in only) (Experimental): Metformin will be given to participants incrementally during a 2 week run in period such that they will receive the clinical dose (2 grams per day). These participants will not participate in the bed rest portion of the protocol.
  Interventions: Drug: Metformin (2 week run-in only)
- Placebo (2 week run-in only) (Placebo Comparator): Placebo will be given to participants incrementally during a 2 week run in period such that they will receive the same amount of pills as the experimental group. These participants will not participate in the bed rest portion of the protocol.
  Interventions: Drug: Placebo (2 week run-in only)

INTERVENTIONS:
Drug: Metformin (Bed Rest) — A clinical oral dose of Metformin will be given to participant daily during bed rest
  Other Names: Metformin hydrochloride; Fortamet; glucophage; Glumetza; Riomet
  Arms: Metformin (Bed Rest)
Drug: Placebo (Bed Rest) — Placebo-comparator. The same quantity of non-active tablets will be given at the same time of day as the Metformin treatment group
  Arms: Placebo (Bed Rest)
Drug: Metformin (2 week run-in only) — A clinical oral dose of Metformin will be given to participant daily during a two week run-in period only.
  Other Names: Metformin hydrochloride; Fortamet; Glucophage; Glumetza; Riomet
  Arms: Metformin (2 week run-in only)
Drug: Placebo (2 week run-in only) — Placebo-comparator. The same quantity of non-active tablets will be given at the same time of day as the Metformin 2 week run-in treatment group.
  Arms: Placebo (2 week run-in only)

SUMMARY:
Muscle atrophy and insulin resistance are common after bed rest in healthy older adults. Metformin treatment has been shown to improve insulin sensitivity and attenuate muscle loss in insulin resistance adults though the mechanisms are not fully known. Metformin used as a preventive strategy to maintain muscle and metabolic health in bed ridden older adults has not been investigated.

DETAILED DESCRIPTION:
Hospitalizations for disease, injury, and/or surgery in older adults are likely to impair physical mobility and, therefore, the older adults capacity to be physically active both during hospitalization and beyond. The resulting sedentary lifestyle is likely to be accepted as the "new normal", ultimately increasing the risk of skeletal muscle and metabolic dysfunction (e.g. insulin resistance and sarcopenia).

Muscle atrophy and insulin resistance are an unfortunate consequence with disuse in older adults. We have observed with our bed rest studies in healthy older adults that in addition to muscle and metabolic changes, we notice increased skeletal muscle inflammation, impaired glucose uptake signaling and an upregulation of enzymes related to de novo ceramide biosynthesis. The accumulation of ceramide, a toxic lipid intermediate, can disrupt glucose homeostasis and impair muscle growth. Metformin treatment has been shown to improve insulin sensitivity and attenuate muscle loss in insulin resistant adults through a mechanism that may involve ceramide synthesis. Metformin used as a preventive strategy to maintain muscle and metabolic health during a period of physical inactivity in older adults has not been investigated.

A separate group of participants for the 2-week Metformin Run-in Period, independent of the bed rest and recovery study will also be recruited. All study procedures will be the same as the 2-week Run-In period within the full protocol.

We hypothesize that metformin treatment in healthy older adults during bed rest would attenuate inflammation, insulin resistance, and thigh muscle loss and changes in lipid accumulating in muscle. We also hypothesize that elevated skeletal muscle ceramide levels, is central to the development of insulin resistance with bed rest in older adults.

Therefore, we have proposed to conduct a clinical study in older adults to:

1. Test if daily metformin treatment (vs placebo) during 5d of bed rest in older adults would attenuate intramuscular ceramide accumulation (lipid accumulation), insulin resistance (euglycemic-hyperinsulinemic clamp), and loss in thigh muscle lean mass. We would also like to determine if 5-days of bed rest in older adults within the placebo group increases skeletal muscle ceramide concentrations and whether these are in turn associated with insulin resistance.
2. Test if daily metformin treatment (vs placebo) during 5d of bed rest in older adults would improve skeletal muscle glucose uptake cell signaling, reduce skeletal muscle inflammation and ceramide biosynthesis signaling.
3. Determine if muscle ceramides and insulin resistance return to baseline levels following 7 days of recovery after bed rest in the placebo group.
4. Determine if metformin given over a 2 week period (independent of bed rest) will improve muscle size, strength and insulin sensitivity.
5. Determine if metformin improves the recovery of muscle size and strength and insulin sensitivity 7 days after bed rest.

These findings will be foundational for future development of treatments to prevent insulin resistance and muscle atrophy in inactive older adults.

ELIGIBILITY:
Inclusion Criteria:

* Age 60y and older
* Ability to sign informed consent
* Free-living, prior to admission

Exclusion Criteria:

* Personal history of cardiovascular disease
* Uncontrolled endocrine or metabolic disease (e.g., hypo/hyperthyroidism, HbA1c ≥6.5%)
* Evidence of kidney disease or failure (defined as serum creatinine > 1.5mg/dL)
* Vascular disease or risk factors of peripheral atherosclerosis. (e.g., uncontrolled hypertension, obesity, diabetes)
* Risk of Deep vein thrombosis including family history of thrombophilia, Deep vein thrombosis, pulmonary emboli, myeloproliferative diseases including polycythemia (Hb>18 g/dL) or thrombocytosis (platelets>400x103/mL)
* Use of anticoagulant therapy (e.g., Coumadin, heparin)
* Uncontrolled hypertension (e.g. systolic pressure >160 or a diastolic blood pressure > 100)
* Cancer or history of successfully treated cancer (less than 1 year) other than basal cell carcinoma
* Currently on a weight-loss diet or body mass index > 30 kg/m2
* Inability to abstain from smoking for duration of study
* HIV or hepatitis B or C*

  * Subjects excluded due to positive screening results, including HIV, hepatitis B or hepatitis C, will be immediately scheduled for counseling and follow-up testing as needed, and will be advised to consult their primary physician.
* Chronic systemic corticosteroid use (≥ 2 weeks) within 4 weeks of enrollment and for study duration (intra-articular/topical/inhaled therapeutic or physiologic doses of corticosteroids are permitted). Androgens or growth hormone within 6 months of enrollment and for study duration (topical physiologic androgen replacement is permitted)
* Subjects with hemoglobin or hematocrit lower than accepted lab values
* History of stroke with motor disability
* A recent history (<12 months) of GI bleed
* Depression [>5 on the 15 items Geriatric Depression Scale (GDS)]*

  *This criteria will only apply to subjects in the bed rest arm.
* Liver disease (the ratio of serum aspartate aminotransferase to serum alanine aminotransferase 2 times above the normal limit, hyperbilirubinemia) History of respiratory disease
* Currently taking estrogen products (topical vaginal products are not exclusionary (e.g. cream))
* Recent travel history as defined by 4 hours of travel by airplane in the last week
* Any other condition or event considered exclusionary by the PI and faculty physician

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Muscle size | Change in muscle size from baseline to 5-days of bed rest will be compared between groups after 5 days of bed rest
  Change in muscle size from baseline to 5-days of bed rest (determined from MRI)
Insulin sensitivity | Change in insulin sensitivity from baseline to 5-days of bed rest will be compared between groups after 5 days of bed rest
  Change in insulin sensitivity from baseline to 5-days of bed rest (determined from glucose infusion rate)

CONTACTS AND LOCATIONS:
Overall Officials: Micah Drummond, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Petrocelli JJ, McKenzie AI, de Hart NMMP, Reidy PT, Mahmassani ZS, Keeble AR, Kaput KL, Wahl MP, Rondina MT, Marcus RL, Welt CK, Holland WL, Funai K, Fry CS, Drummond MJ. Disuse-induced muscle fibrosis, cellular senescence, and senescence-associated secretory phenotype in older adults are alleviated during re-ambulation with metformin pre-treatment. Aging Cell. 2023 Nov;22(11):e13936. doi: 10.1111/acel.13936. Epub 2023 Jul 24. PMID 37486024
- [Derived] Petrocelli JJ, de Hart NMMP, Lang MJ, Yee EM, Ferrara PJ, Fix DK, Chaix A, Funai K, Drummond MJ. Cellular senescence and disrupted proteostasis induced by myotube atrophy are prevented with low-dose metformin and leucine cocktail. Aging (Albany NY). 2023 Mar 20;15(6):1808-1832. doi: 10.18632/aging.204600. Epub 2023 Mar 20. PMID 36947713
- [Derived] McKenzie AI, Mahmassani ZS, Petrocelli JJ, de Hart NMMP, Fix DK, Ferrara PJ, LaStayo PC, Marcus RL, Rondina MT, Summers SA, Johnson JM, Trinity JD, Funai K, Drummond MJ. Short-term exposure to a clinical dose of metformin increases skeletal muscle mitochondrial H2O2 emission and production in healthy, older adults: A randomized controlled trial. Exp Gerontol. 2022 Jun 15;163:111804. doi: 10.1016/j.exger.2022.111804. Epub 2022 Apr 9. PMID 35405248